CLINICAL TRIAL: NCT02632890
Title: Evaluation of the Effectiveness of the Abatacept (Orencia®) IV and SC Patient Alert Cards in Patients With Rheumatoid Arthritis in European Economic Area Countries
Brief Title: Assessment of the Effectiveness of IV and SC Abatacept (Orencia) Patient Alert Cards in Patients With Rheumatoid Arthritis in a Sample of EU Countries
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-537
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients survey: Adult patients treated with abatacept for rheumatoid arthritis
- HCP survey: HCP with at least 1 patient taking abatacept
- Retrospective chart review study: Adult patients treated with abatacept for rheumatoid arthritis

SUMMARY:
The purpose of the study is to determine a) if the implementation of abatacept (Orencia®) patient alert card (PAC) resulted in effective understanding of key safety messages and b) if the degree of understanding of key safety messages is associated with improved clinical and safety outcomes.

DETAILED DESCRIPTION:
3 sub studies: 2 Cross-Sectional and 1 retrospective chart review

ELIGIBILITY:
Inclusion Criteria:

* Patient survey (cohort 1):

  1. Patients has taken abatacept within the previous 3 months for rheumatoid arthritis
  2. Patient is 18 years of age or over
* HCP survey (cohort 2):

  a) Physician or nurses working in rheumatology centers, with at least 1 patient taking abatacept in the previous 6 months for rheumatoid arthritis (by prescribing, administering or by follow up)
* Retrospective chart review study (cohort 3):

  1. Patient survey questionnaire completed , Informed Consent Form (ICF) signed

Exclusion Criteria:

* Patient survey:

  1. Patient has participated in a clinical trial for their arthritis in the previous 12 months
  2. Currently an employee of BMS
* HCP survey:

  1. Physicians or nurse who have recruited patients for the Patient survey
  2. Currently an employee of BMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Patients enrolled by physician or nurse based in hospital rheumatology departments and physician clinics and offices
  Cohort 2: Physician or nurse based in hospital RA department and physician clinics and offices
  Cohort 3: Patients enrolled by physician or nurse based in hospital rheumatology departments and physician clinics and offices
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Patient survey: Proportion of patients treated with abatacept who are aware of the existence of the PAC | At patient enrolment
Patient survey: Proportion of patients treated with abatacept who have received the PAC | At patient enrolment
Patient survey: Proportion of patients who have utilised the PAC, and the extent of its use | At patient enrolment
Patient survey: Levels of patient knowledge and comprehension related to the important identified risks of allergic reactions associated with abatacept treatment | At patient enrolment
Patient survey: Levels of patient knowledge and comprehension related to the important identified risks of associated with abatacept treatment | At patient enrolment
Patient survey: Mean scores for correct responses for questions grouped by objectives | At patient enrolment
  Objectives: distribution, awareness, utility, utilization and knowledge
Patient survey: Mean total score for correct responses | At patient enrolment
HCP survey: Proportion of HCPs who prescribe or administer abatacept in rheumatology centers who are aware of the PAC | Day 1
HCP survey: Proportion of HCPs' who have utilized the PAC, and the extent of its use | Day 1
HCP survey: Levels of HCPs' knowledge and comprehension related to the important identified risks of infections and the need to screen for specific infection prior to initiating or administering abatacept | Day 1
HCP survey: Mean total score for correct responses | Day 1
HCP survey: Mean scores for correct responses for questions grouped by objectives | Day 1
  Objectives: distribution, awareness, utility, utilization and knowledge
Retrospective chart review study (clinical outcome study): Proportion of infections leading to hospitalization | Approximately 3 months

SECONDARY OUTCOMES:
Major determinants of patients knowledge of the key messages contained in the abatacept IV, Subcutaneous (SC) formulation PACs among patients | At patient enrolment
  Determinants: Formulation of abatacept administered, country, age, gender,
  educational level, duration of arthritis, number of prescription medications, duration of therapy with abatacept, HCP guided or self-administration
Major determinants of understanding the key messages contained in the abatacept IV, SC formulation PACs among patients | At patient enrolment
  Determinants: Formulation of abatacept administered, country, age, gender,
  educational level, duration of arthritis, number of prescription medications, duration of therapy with abatacept, HCP guided or self-administration
Major determinants of implementation regarding the key messages contained in the abatacept IV, SC formulation PACs among patients | At patient enrolment
  Determinants: Formulation of abatacept administered, country, age, gender,
  educational level, duration of arthritis, number of prescription medications, duration of therapy with abatacept, HCP guided or self-administration
Determinants of Health Care Professional (HCP) understanding, Implementation regarding key messages contained in the PAC based on data collected in the abatacept IV and SC formulation PACs among HCPs | Day 1
  Determinants: type of HCP, role of the HCP, country, age and sex of the HCP, years in the specialty, number of HCPs in the unit, annual number of patients managed by the unit, number of patients for whom abatacept was prescribed in the previous 12 months, type of practice, type of institution (academic or non-academic), size of town
Retrospective chart review study (clinical outcome study): Proportion of patients with results of any test to screen for Tuberculosis (TB) prior to administration of therapy of abatacept | Upto 8 years
Retrospective chart review study (clinical outcome study): Proportion of patients with results of any test to screen for viral hepatitis before administration of therapy with abatacept | Upto 8 years
Retrospective chart review study (clinical outcome study): Mean time from infection (symptom onset) to receiving medical attention | Upto 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- France (2):
  - CHU Limoges - Hopital Dupuytren, Limoges
  - APHM - Hopital Sainte-Marguerite, Marseille, Paris
- Germany (10):
  - Acura Kliniken, Bad Kreuznach
  - Local Institution, Bad Kreuznach
  - Bad Nauheim, Bad Nauheim
  - Local Institution, Bad Nauheim
  - Local Institution, Frankenberg
  - Local Institution, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Heidelberg, Heidelberg
  - Local Institution, Zwickau
  - Zwickau, Zwickau
- Spain (13):
  - Hospital Coruña, A Coruña
  - Hospital Ccal. de Barbastro, Barbastro
  - Hospital Elche, Elche
  - Hospital Elda, Elda
  - Local Institution, Elda
  - Hospital Getafe, Getafe
  - Hospital Gregorio Marañon, Madrid
  - Local Institution, Madrid
  - Hospital Merida, Mérida
  - Hospital Virgen del Puerto, Plasencia
  - Local Institution, Plasencia
  - Hospital Virgen Macarena, Seville
  - Hospital Mutua de Terrasa, Terrassa
- Sweden (2):
  - Local Institution, Malmo
  - Local Institution, Solna
- United Kingdom (9):
  - Nevil Hall Hospital, Abergavenny
  - Local Institution, Basingstoke
  - Royal Derby Hospital, Derby
  - Barnsley Hospital NHS Foundation Trust, Dewsbury
  - Eastbourne District Gen. Hosp., East Sussex
  - Local Institution, Harlow
  - Princess Alexandra Hospital, Harlow
  - Arrow Park Hospital, Metropolitan Borough of Wirral
  - St Helens Hospital, St Helens

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx